CLINICAL TRIAL: NCT03744975
Title: Effects of Neprilysin Inhibition With ARNI (LCZ 696) on the Cardiorenal and Humoral Response to Acute Saline Volume Expansion in DM With and Without PDD
Brief Title: PDD in Type 2 Diabetes w/wo Diastolic Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Horng Chen, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-006589
Record Dates: First submitted 2018-04-19; First posted 2018-11-19 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; Diastolic Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: Placebo-controlled study comparing Oral Placebo with Oral LCZ 696 (Entresto)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebos (Placebo Comparator): Control Intervention will be 1 Placebo Capsule given orally, one time
  Interventions: Drug: Placebos
- LCZ 696 (Active Comparator): 1st Experimental Arm will be 1 capsule of LCZ 696 given orally, one time
  Interventions: Drug: LCZ 696; Drug: Placebos

INTERVENTIONS:
Drug: LCZ 696 — Participants will receive Oral LCZ 696 (Entresto 97/103 mg)
  Other Names: Entresto®); ARNI
  Arms: LCZ 696
Drug: Placebos — Participants will receive 1oral Placebo capsule
  Other Names: Placebo capsule

SUMMARY:
This study will advance the investigator's knowledge of the integrated cardiorenal and humoral physiology in type 2 diabetic patients with and without pre-clinical diastolic dysfunction, and test a novel therapeutic strategy which may prevent a progression to symptomatic Stage C heart failure

DETAILED DESCRIPTION:
6.1 Visit 1 Consent Visit: Possible study participants will meet with study coordinator to review consent form. After enrollment into the study, a 6-minute walk will be performed (minimum required distance: 450 meters). Diet instructions will be given by a dietician about a no added salt diet, 120 mEq Na/day, which will be maintained throughout the study period. Comprehensive metabolic panel (including albumin, bilirubin, calcium, bicarbonate, chloride, creatinine, glucose, alkaline phosphatase, potassium, total protein, sodium, AST, ALT and BUN)and complete blood count with differential will be obtained. Brief physical exam or nursing assessment will be performed by a qualified Study Team Member. Visit 2 will be scheduled at least one week out from consent visit to accommodate diet compliance, unless participant is already compliant with salt intake parameter. Instructions for completing a 24-hour urine collection, and container for Study Visit 2, will be given.

Subjects who are taking angiotensin converting enzyme inhibitors (ACEI) will be switched over to an equivalent dose of Valsartan or Losartan, which will be maintained for 3 days beyond the end of the study period. This is due to the FDA recommendation that patients on ACEI should have a 36 hour washout period before administering ARNI due to the increased risk of angioedema.

6.2 Visit 2 Participants will start a twenty-four hour urine collection one day prior to the active study day for assessment of baseline sodium excretion, creatinine clearance and urine protein analysis.

Subjects will be admitted to the Clinical Research Translational Unit (CRTU). On the active study day, subjects will withhold their usual dose of medications and will be placed in the supine position for 1 hour. During the first 15 minutes, two standard intravenous (IV) catheters will be placed (one in each arm). One catheter will be used for infusion and the other (in the contralateral arm) for blood sampling. A bladder ultrasound will be completed after the participant's first void after admitting to assess for urine retention. Subjects will be asked to drink 10ml/Kg of water to insure sufficient urinary flow. A priming dose (calculated according to body size) of Iothalamate, to measure glomerular filtration rate (GFR), is infused, followed by a constant rate IV sustaining dose (calculated according to estimated kidney function) of Iothalamate. The subjects will be asked to empty their bladder spontaneously every thirty minutes (if subjects are unable to void every thirty minutes, a urinary catheter will be used upon consent). Throughout the study, at the end of each 30-minute clearance period, subjects will be asked to drink an amount of water equivalent to the sum of the blood losses and the urinary flow.

After an equilibration period of 45 minutes, a 30-minute baseline renal clearance will be carried out. Urinary samples for determination of volume, urinary sodium excretion (UNaV), cGMP, and Iothalamate will be obtained at the end of the clearance period. Venous blood samples for Iothalamate, sodium, ANP, BNP, cGMP, soluble neprilysin, renin, angiotensin II and aldosterone will be obtained at the middle of the clearance period. Blood pressure will be measured at 20-minute intervals by using an automatic blood pressure cuff, and heart rate will be continuously monitored by electrocardiography. Echocardiography will be performed during these baseline clearances to determine left atrial (LA) and LV volumes and systolic and diastolic function.

After the baseline clearance, the subjects will be randomized to receive either a) oral placebo or b) Oral ARNI (LCZ 696/Entresto 97/103 mg). Previous studies have demonstrated that the maximum effect for LCZ 696 is about 1.5 hours after oral administration. Hence, one and one-half hours after the administration of the oral medication, the acute saline load will be administered (normal saline 0.9% 0.25 ml/kg/min for 1 hour). Two 30-minute clearances (as outlined above) will be repeated with the subjects in a supine position during the saline infusion. As above, blood samples are collected midway during each clearance and urine samples are obtained every 30 minutes. Echocardiography will be repeated immediately after the end of the saline infusion, after which subjects will be allowed to eat a meal and be dismissed.

The subjects will return after at least 1 week of washout for the second crossover study. Container for 24-hour urine collection for Study Visit 3 will be given.

6.3 Visit 3 Visit 3 will take place the same as described in Visit 2, receiving one of the 2 medication administrations not received on Visit 2: (a) oral placebo or b) Oral ARNI (LCZ 696/Entresto 97/103 mg)).

At the end of Visit 3, study participation is complete.

ELIGIBILITY:
Inclusion Criteria

* Type 2 diabetes mellitus
* On at least one oral hypoglycemic agent, or glucagon-like peptide analogue or insulin, for at least 6 months
* EF > 50% without diastolic dysfunction or EF > 50% with grade 2 or more diastolic dysfunction, without prior diagnosis, or signs and symptoms, of heart failure
* Minimal distance of >450 meters on a 6-minute walk. If the subject is not able to walk 450 meters due to pain in hips and/or knees, and not fatigue or shortness of breath, then they will still qualify for the protocol.

Exclusion Criteria

* HbA1C> 9 % at enrollment
* prior diagnosis, or signs and symptoms, of heart failure;
* Currently taking a loop diuretic
* myocardial infarction within 6 months of Visit 2
* unstable angina within 6 months of Visit 2
* significant (> moderate) valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis
* severe congenital heart diseases
* sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
* second or third degree heart block without a permanent cardiac pacemaker
* stroke within 3 months of screening, or other evidence of significantly compromised CNS perfusion
* ALT >2 times the upper limit of normal
* serum sodium of < 125 mEq/dL or > 160 mEq/dL
* serum potassium of < 3.5 mEq/dL or > 5.9 mEq/dL
* hemoglobin < 9 gm/dl
* eGFR < 30 ml/min (at screening)
* other acute or chronic medical conditions or laboratory abnormality which may increase the risks associated with study participation or may interfere with interpretation of the data
* received an investigational drug within 1 month prior to dosing;
* patients with an allergy to iodine
* female subject who is pregnant or breastfeeding
* in the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Plasma cGMP Response | 3 months
  The change in plasma cGMP levels from baseline to after volume expansion DM with PDD versus non-PDD

SECONDARY OUTCOMES:
Renal response | 3months
  The composite endpoint consisting of sodium excretion, GFR, urinary cGMP and diastolic function change from baseline to volume expansion in Type 2 DM with PDD versus non-PDD

CONTACTS AND LOCATIONS:
Overall Officials: Horng H Chen, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No